CLINICAL TRIAL: NCT04035837
Title: A Study of Peg-interferon Treatment for Nucleos(t)Ide Analogues Suppressed Chronic Hepatitis B Patients With Low Level Hepatitis Surface Antigen
Brief Title: The Clinical Cure Project of Chronic Hepatitis B in China
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhiliang Gao, The director of the infectious diseases department, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZhuFeng Project
Record Dates: First submitted 2019-07-13; First posted 2019-07-29 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- short-course combination group (Experimental): Nucleoside analogue is used during the first 3 months.
  Interventions: Drug: pegylated interferon-alfa
- full-course combination group (Experimental): Nucleoside analogue is used during all the course of study.
  Interventions: Drug: pegylated interferon-alfa
- Monotherapy group (Experimental): Only Peg-IFN is used during all the course of study.
  Interventions: Drug: pegylated interferon-alfa

INTERVENTIONS:
Drug: pegylated interferon-alfa — All the patients in this study will receive pegylated interferon for all course.

SUMMARY:
Chronic hepatitis B is a global public health problem, with nearly 700,000 deaths each year because of hepatitis B-related diseases. Recent studies have found that some patients who have used nucleot(s)ide analogues(NAs) for some period can achieve higher hepatitis B surface antigen(HBsAg) clearance rate(which is called clinical cure or functional cure) by using pegylated interferon. Patients who achieve clinical cure will further reduce liver inflammation, fibrosis and risks of liver cirrhosis and cancer in the future. This study was initiated in May 2018 and plans to recruit 30,000 eligible patients. The enrollment conditions are as follows: 1. according with the diagnosis of chronic hepatitis B in the guideline of China in 2015; 2.18-60 years old; 3. more than 1 year history of NAs therapy with HBsAg ≤1500 IU/ml, negative hepatitis e antigen and hepatitis B virus DNA<100 IU/ml; 4. no contraindications of interferon. For the above patients, pegylated interferon was used for 1-2 years(combined with NAs for at least 3 months).The primary goal of this study is to find out the optimal treatment for clinical cure.

ELIGIBILITY:
Inclusion Criteria:

* according with the diagnosis of chronic hepatitis B in the guideline of China in 2015
* 18-60 years old
* more than 1 year history of nucleot(s)ide analogues therapy with HBsAg ≤1500 IU/ml, negative HBeAg and HBV DNA<100 IU/ml
* no contraindications of interferon

Exclusion Criteria:

* Allergy to interferon
* Alanine transaminase >10 times of upper limit of normal(ULN) or total bilirubin >2 times of ULN
* existing or previous decompensated liver cirrhosis
* White blood cells or Platelet below the lower limit of normal
* existing severe organ injury
* combined with autoimmune diseases, psychiatric diseases, diabetes or thyroidism
* confirmed or suspected malignant tumors
* before or after transplantation
* using immunosuppressor
* pregnant or having a planned parenthood in 2 years
* alcohol or drug addicted
* infected by HIV
* any conditions that is unsuitable to interferon therapy according to the doctors' judgement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30000 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
hepatitis B surface antigen | up to 48 weeks
  hepatitis B surface antigen should be tested by the reagents from Roche or Abbott, which is expressed by using IU/ml.

SECONDARY OUTCOMES:
hepatitis B surface antibody | up to 48 weeks
  hepatitis B surface antigen should be tested by the reagents from Roche or Abbott, which is expressed by using IU/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiliang Gao, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Department of Infectious Diseases, The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Study protocol would be shared with other researchers.

REFERENCES:
- [Background] Fattovich G, Bortolotti F, Donato F. Natural history of chronic hepatitis B: special emphasis on disease progression and prognostic factors. J Hepatol. 2008 Feb;48(2):335-52. doi: 10.1016/j.jhep.2007.11.011. Epub 2007 Dec 4. PMID 18096267
- [Background] Liaw YF, Chu CM. Hepatitis B virus infection. Lancet. 2009 Feb 14;373(9663):582-92. doi: 10.1016/S0140-6736(09)60207-5. PMID 19217993
- [Background] Brunetto MR. A new role for an old marker, HBsAg. J Hepatol. 2010 Apr;52(4):475-7. doi: 10.1016/j.jhep.2009.12.020. Epub 2010 Jan 30. No abstract available. PMID 20185190
- [Background] Liu J, Lee MH, Batrla-Utermann R, Jen CL, Iloeje UH, Lu SN, Wang LY, You SL, Hsiao CK, Yang HI, Chen CJ. A predictive scoring system for the seroclearance of HBsAg in HBeAg-seronegative chronic hepatitis B patients with genotype B or C infection. J Hepatol. 2013 May;58(5):853-60. doi: 10.1016/j.jhep.2012.12.006. Epub 2012 Dec 13. PMID 23246508
- [Background] Tseng TC, Liu CJ, Su TH, Wang CC, Chen CL, Chen PJ, Chen DS, Kao JH. Serum hepatitis B surface antigen levels predict surface antigen loss in hepatitis B e antigen seroconverters. Gastroenterology. 2011 Aug;141(2):517-25, 525.e1-2. doi: 10.1053/j.gastro.2011.04.046. Epub 2011 Apr 28. PMID 21672542
- [Background] Moucari R, Korevaar A, Lada O, Martinot-Peignoux M, Boyer N, Mackiewicz V, Dauvergne A, Cardoso AC, Asselah T, Nicolas-Chanoine MH, Vidaud M, Valla D, Bedossa P, Marcellin P. High rates of HBsAg seroconversion in HBeAg-positive chronic hepatitis B patients responding to interferon: a long-term follow-up study. J Hepatol. 2009 Jun;50(6):1084-92. doi: 10.1016/j.jhep.2009.01.016. Epub 2009 Mar 9. PMID 19376603
- [Background] Dietary effects on diurnal variation in lipogenesis. Nutr Rev. 1987 May;45(5):157-8. doi: 10.1111/j.1753-4887.1987.tb06353.x. No abstract available. PMID 3601258
- [Background] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Background] Thompson AJ, Nguyen T, Iser D, Ayres A, Jackson K, Littlejohn M, Slavin J, Bowden S, Gane EJ, Abbott W, Lau GK, Lewin SR, Visvanathan K, Desmond PV, Locarnini SA. Serum hepatitis B surface antigen and hepatitis B e antigen titers: disease phase influences correlation with viral load and intrahepatic hepatitis B virus markers. Hepatology. 2010 Jun;51(6):1933-44. doi: 10.1002/hep.23571. PMID 20512987
- [Background] Ning Q, Han M, Sun Y, Jiang J, Tan D, Hou J, Tang H, Sheng J, Zhao M. Switching from entecavir to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: a randomised open-label trial (OSST trial). J Hepatol. 2014 Oct;61(4):777-84. doi: 10.1016/j.jhep.2014.05.044. Epub 2014 Jun 7. PMID 24915612
- [Derived] Chang LJ, Hao CQ, Rao GR, Xu LL, Li J, Cheng Y, Zheng LJ, Wu CW, Chen HX, Chen ZR, Lian JQ, Wu SH, Luo LM, Zhang WL, Zhang Y. Recurrence risk factors for chronic hepatitis B virus-infected patients who achieve functional cure with pegylated interferon-alpha-2b-based therapy: a multicenter pilot study. Virol J. 2025 May 19;22(1):146. doi: 10.1186/s12985-025-02761-3. PMID 40390028
- [Derived] Wang Z, Wang X, Zhou L, Shi S, Hua Y, Feng Y. Safety and efficacy of 48-week pegylated interferon-alpha-2b therapy in patients with hepatitis B virus-related compensated liver cirrhosis: a pilot observational study. Front Med (Lausanne). 2024 Dec 4;11:1489671. doi: 10.3389/fmed.2024.1489671. eCollection 2024. PMID 39697201
- [Derived] Huang Q, Xiao X, Zhuang X, Chen W, Huang Y, Liao J, Wang W, Wang Y, Lu L, Liu Z, Huang J. Peripheral Circulating Exosomal-miRNAs Potentially Mediate the Sensitivity to Interferon Treatment in Chronic Hepatitis B Virus Patients. Viral Immunol. 2023 Apr;36(3):209-221. doi: 10.1089/vim.2022.0130. Epub 2023 Mar 21. PMID 36944116